CLINICAL TRIAL: NCT01587157
Title: Capnography During Percutaneous Transhepatic Cholangiodrainage (PTCD) (HepaBreath)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Prevention
Other Study IDs: 20042012
Record Dates: First submitted 2012-04-23; First posted 2012-04-30 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Apnea; Hypoxemia; Complications
MeSH Terms: conditions — Apnea; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- capnography (Experimental)
  Interventions: Procedure: capnography

INTERVENTIONS:
Procedure: capnography

SUMMARY:
Capnography provides noninvasive monitoring of ventilation and can allow early recognition of altered respiration patterns and apnea. The aim of this prospective study was to compare the detection of apnea and the prediction of oxygen desaturation and hypoxemia by capnography versus clinical surveillance during procedural sedation for percutaneous transhepatic cholangiodrainage (PTCD).

ELIGIBILITY:
Inclusion Criteria:

* Age>=18
* Scheduled for PTCD with midazolam and propofol sedation

Exclusion Criteria:

* age less than 18 years
* ASA class V
* allergy to narcotic drugs
* pregnancy
* pre-existing hypotension, bradycardia or hypoxemia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
mean cumulative duration of detected apnea episodes per patient (capnographic vs. clinical surveillance)

SECONDARY OUTCOMES:
overall number of detected episodes of apnea
the occurrences of oxygen desaturation and hypoxemia

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum rechts der Isar, Munich, Bavaria, Germany